CLINICAL TRIAL: NCT03082521
Title: Better Antibiotic Prescribing Through Action Research
Acronym: BAbAR
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Annelies Colliers, Principal Investigator, Universiteit Antwerpen
Other Study IDs: BAbAR
Record Dates: First submitted 2017-03-07; First posted 2017-03-17 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Infectious Disease
Keywords: After hours care; Primary care; Antibiotics; Action Research
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Improving the antibiotic prescribing quality — The goal is to improve the antibiotic prescribing quality of GPs in a GPC by setting up a participatory action research. The interventions will be co-designed with the GPs.

SUMMARY:
This PAR (participatory action research) study to improve antibiotic prescribing quality in a GPC (general practitioner cooperative) during OOH-care (out-of-hours-care) uses a mixed methods approach using qualitative as well as quantitative techniques. In a first exploratory phase we will work on partnership development and mapping the existing issues. In a second phase the focus will be on facilitating change and implementing interventions through PDSA (plan do study act) cycles. In a third phase outcomes on prescribing quality during and outside office hours will be evaluated. Equally important is the process evaluation and theory building on improving antibiotic prescribing through PAR.

DETAILED DESCRIPTION:
Phase 1: Exploring In the exploratory phase of this research the focus will first be on partnership development and engaging the GPs with this research project. The success of the PAR approach depends on the willingness of the stakeholders to play an active role.

To map the willingness to participation and the need to change, contacts with the GPs of the GPC are planned. Emphasis will be put on the fact that the partnership is non-judgmental, has a reciprocal character, and is based on trustworthiness. Developing a positive partnership with the GPs will be essential. A first contact with the board of the GPC has already taken place, and they expressed their willingness to participate in this project.

Next, narrative research will be undertaken to explore how the different stakeholders experience or make sense of antibiotic prescribing within their setting. By better understanding GPs' behaviour and taking into account the different barriers they experience, we will be able to understand their conduct and to develop interventions with better chances of success and bigger support from the GPs. Individual in-depth interviews will be performed with the relevant identified stakeholders (GPs, manager, etc.). A semi-structured interview guide will be used. Topics consist on the one hand on the specifics on prescribing antibiotics in OOH primary care, the perceived need and the receptiveness to change, local antibiotic prescribing culture and habits etc. and on the other hand on the willingness to participate in PAR, the degree of commitment in being a co-researcher, the perceived viability of the project etc. Purposeful sampling will be performed to obtain a relevant variety in participants that reflects our specific setting (young vs experienced GPs, solo vs group practice during office hours, ethnical background etc.). Scientific rigour is ensured by using triangulation and member checks involving first the participants in the interviews and second all other stakeholders (see Phase 2). The GPs who have contributed to the interviews will receive a formal analysis report with the summary of the findings and will be asked to deliver feedback (member checking, but also reflecting on it) in a focus group. In a second phase this will be made available to all GPs of the GPC. Coding of the first three to five interviews will be done by two researchers independently (AC, a GP and SA, a sociologist). The coding framework will then be developed by consensus of these two researchers. Following the independent coding, the initial thematic framework will be compared, and similarities and differences will be discussed and amended to create a set of themes that represents both analyses. This thematic framework will be used for further analysis and if new themes emerge this will be discussed amongst the research team. The interim analyses will be critically looked at by the other three members of the multidisciplinary research team and will be adapted after their feedback.

To develop a clear view on the why and when antibiotics are prescribed in OOH primary care an ethnographic study will be setup. If consent is given by the GPs we will use video observations to achieve a better understanding of the context, difficulties, clinical issues, patient-doctor interactions etc. during prescribing antibiotics in OOH primary care. It gives the possibility to gain insight in GPs habits in their natural, real-world setting. The videos will be observed solely by the research team. Complete anonymity of the GPs and patients will be guaranteed. Using video-observations can be a sensitive method for GPs in practice, but a review showed that from an ethical and practical point of view recording consultations is generally acceptable to both patients and GPs. The data collected through video observations will be analysed on the one hand for research purposes and on the other hand to guide the intervention development. During the interviews of phase 1 the use of video-observations and possible related barriers will be discussed with the participants. During the interviews we explore the thoughts of the GPs about receiving personal feedback or the possibility to discuss the videos with one of the researchers or with their peers. Another question is asked about the thoughts about using the videos solely as transcripts for research or also for peer education, or even to use them in video-format with peers. Hence, the way we will use the video material will depend on the willingness or preference of the participants in our action research.

Because PAR is setup together with the participants having a voice in the design of the study, alternative data collection methods to gain insight in the daily practice of using antibiotics in OOH primary care can be suggested and subsequently applied. Alternative methods could be a live observation by a member of the research team, a study of the anonymised electronical medical health records, standardised patients, patient interviews, case vignettes, etc..

Antibiotic prescribing quality at the level of the GPC will be assessed before the start of the PAR using well-established APQI applied before in this setting. For the six most common indications for antibiotic prescribing (in descending order: acute bronchitis (ICPC (6) code R78), acute upper RTI (R74), cystitis/other urinary infection (UTI; U71), acute tonsillitis (R76), acute/chronic sinusitis (R75), and acute otitis media (H71)) and for pneumonia (R81) values of three quality indicators will be calculated and fed back:

1. = the percentage of patients prescribed an antibiotic;
2. = a. and receiving the guideline recommended antibiotic;
3. = a and receiving quinolones. The APQI values will be calculated before the start of the PAR in phase 1 and will be used during the PDSA (plan-do-study-act) cycle(s) of phase 2 as a quantitative indicator of antibiotic prescribing quality improvement in OOH primary care. In the data-analyses the focus will be on lowering antibiotic prescribing as well as on improving the proportion of receiving a recommended antibiotic and lowering the use of broad-spectrum antibiotics. But, the involved GPs can choose to develop interventions that target all these elements or target only one specific problem. The participants will have their saying not only in the action process itself, but also on how it will be evaluated so matching interventions and assessments have to be chosen.

We will be able to use data collected through the electronic medical health records. iCAREdata (Improving Care And Research Electronic Data Trust Antwerp; www.icaredata.eu), i.e. a research database linking and collecting routine data from all GPCs covering out-of-hours primary care in Antwerp, allows us to deliver up to date feedback and evaluate interventions at GPC level.

Phase 2: Facilitating change Next PAR will focus on planning and implementing interventions, based on the findings in phase 1. Participants are encouraged to be involved in defining the nature of change and the activities to accomplish this change.

In the second phase of our study qualitative and quantitative results of phase 1 will be fed back to all participants in the PAR. In reflective peer group sessions the barriers and opportunities will be explored and interventions will be co-designed together with PAR participants taking into account previous work as well as the current scientific knowledge. By reflecting and interacting with each other, a joint strategy grounded in the reality of OOH primary care practice can originate. Interventions will be delivered and assessed at GPC level, but since the intervention(s) will be co-created with the stakeholders, at this stage it is unclear how the intervention will look like and at who it will be aimed, the individual GP, the patients, both or any other relevant stakeholder or structure. Every GP of the region is on call for several times every year and thus will be exposed to the intervention(s). There are recognised difficulties in measuring effectiveness of interventions in PAR and using PDSA cycles, because of the many variables in a complex situation. The evaluation of action research therefore is not solely a change intervention, but more a research approach with change and knowledge outcomes, where qualitative findings on context, process and views of participants are a part of.

The feasibility and acceptability of the implemented interventions will be studied from the perspectives of the GPs, but also from the perspective of the patients. Process indicators will depend on the type of interventions and implementation strategies chosen by the stakeholders. If, for example, they choose for an internet-based communication skills training such as GRACE INTRO, the number of patient information booklets, which are an integral part of this intervention, distributed to patients could serve as a process indicator. But also the experiences, views, acceptability, etc. of patients receiving this intervention will be explored and be taken into account into the adaptation of the interventions. At this point the research group does not have a preference for the type of interventions that will be implemented, but they do have the knowledge of existing, appropriate and effective interventions to support the GPs wishes and needs. We aim to run the PDSA cycle a minimum of two times.

The results of this implementation phase of the study will be reported using the "Standards for Reporting Implementation Studies" (StaRI) checklist.

Phase 3: Evaluation In the third phase the impact of the interventions on the quality of antibiotic prescribing will be evaluated. But equal importance will be given to the evaluation of the process of PAR.

We will evaluate the quality of antibiotic prescribing based on the APQI values for OOH primary care, but also aim to assess any spill over effect to primary care during office hours of improving the quality of antibiotic use outside office hours. The effect on antibiotic use during office hours will be assessed using Intermutualistic Agency (IMA, www.nic-ima.be) data. Hence, the latter outcome measurement will have complete response, and will not interfere with the normal routine of the eligible GPs, allowing a more valid estimate of any spill over effect than databases who recover data from the recording by GPs into their own system. Since IMA data have no link with diagnoses and are data from the dispensing of the medication to the patient, the effect on antibiotic use in general and in relevant subgroups defined by age and gender will be assessed rather than the prescribing by diagnosis. The quality of the IMA data does not depend on the quality of recording by the GPs, in contrast to the OOH care data. In Belgium every GP is obliged to be on call in the GPC of his/her own region, meaning that one GPC covers all the GPs of one specific well-defined region.

The process evaluation aims to deepen our understanding of how, why and what was learnt from the project. Participatory Action Research refers to a range of research methods that emphasise the importance of participants and action. It uses methods that involve iterative processes of reflection and action. Although most of the PAR methods involve qualitative techniques, increasingly quantitative and mixed methods are used, which we will also combine. The main emphasis however is on the process. The main objectives are to explore, to see whether the process is adequate (to see whether the intervention and outcomes are occurring (so is there a change in prescribing)) and to explain how and why does implementation of the intervention lead to effects (so develop or expand a theory to explain the relationships between concepts and the reason for the change).The concept of analytic generalisation, by linking our particular findings to theory, allows to apply the research findings not only in similar contexts, but to other groups and contexts as well.45 Dissemination of this model to other GPCs and other GP settings is one of the deliverables.

ELIGIBILITY:
Inclusion Criteria:

* GPs working in the GPC

Exclusion Criteria:

* /

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General practitioners within a general practitioner cooperative during out-of-hours care.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Interview study | year 1
  Semi-structured interview with the stakeholders on the experiences of prescribing antibiotics in OOH care and the willingness to participate in PAR.
Antibiotic prescribing feedback using antibiotic prescribing quality indicators | year 1
  Using antibiotic prescribing quality indicators (APQI) feedback on the antibiotic prescription rates of the GPC will be generated. For the six most common indications for antibiotic prescribing (in descending order: acute bronchitis (ICPC (6) code R78), acute upper RTI (R74), cystitis/other urinary infection (UTI; U71), acute tonsillitis (R76), acute/chronic sinusitis (R75), and acute otitis media (H71)) and for pneumonia (R81) values of three valid antibiotic prescribing quality indicators (APQI)quality indicators will be calculated and fed back: (5)
  1. = the percentage of patients with age and/or gender limitation prescribed an antibiotic;
  2. = a. and receiving the guideline recommended antibiotic;
  3. = a and receiving quinolones.
Ethnographic study: explanatory and descriptive approach of observations, descriptions and interpretation of the phenomenon of prescribing antibiotics in OOH care | year 2
  Observations of consultations to get a better understanding of the context , difficulties, clinical issues, etc. of prescribing antibiotics in OOH care.
Focus groups (descriptative & interpretative) & description of PDSA cycles on developing and implementing interventions on antibiotic prescribing in OOH care | year 3
  Qualitative and quantitative results of phase 1 will be fedback to the group of GPs. In reflective peer group sessions the issues and problems will be explored and interventions will be designed taking into account previous work.
  The implemented interventions and changes will be studied based on both outcome as process indicators. ESACs' Antibiotic Prescribing Quality Indicators (APQI) will be used to assess quality of antibiotic prescribing. Pocess indicators will depend on the chosen interventions.
Process evaluation and sociological meso-theory building of PAR in the case of improving antibiotic prescribing behaviour in a GPC | year 4
  Evaluation of the study, theory building on optimising antibiotic use with PAR. Study of group-level interactions, descriptive.

SECONDARY OUTCOMES:
Use of Antibiotics (quantity, type, use of broad-spectrum antibiotics,etc.) in daytime care | year 5
  The use of antiobiotics during office hours to assess any spill over effect of PAR in OOH-care.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Coenen, MD, PhD, Study Chair — Universiteit Antwerpen; Sibyl Anthierens, PhD, Study Chair — Universiteit Antwerpen
Locations (1):
- GPC Brabo, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colliers A, Coenen S, Remmen R, Philips H, Anthierens S. How do general practitioners and pharmacists experience antibiotic use in out-of-hours primary care? An exploratory qualitative interview study to inform a participatory action research project. BMJ Open. 2018 Sep 28;8(9):e023154. doi: 10.1136/bmjopen-2018-023154. PMID 30269072
- [Derived] Colliers A, Coenen S, Philips H, Remmen R, Anthierens S. Optimising the quality of antibiotic prescribing in out-of-hours primary care in Belgium: a study protocol for an action research project. BMJ Open. 2017 Oct 15;7(10):e017522. doi: 10.1136/bmjopen-2017-017522. PMID 29038184